CLINICAL TRIAL: NCT05792696
Title: Effectiveness of Peripheral Perfusion Index Guided Strategies for the Prevention and Treatment of Hypotension: a Randomized Trial
Brief Title: PPI Guided Strategies for Prevention and Treatment of Intraoperative Hypotension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: zhiqiang zhou (Other)
Responsible Party: Sponsor-Investigator, zhiqiang zhou, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TJ-IRB20230247
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2023-12

CONDITIONS: Intraoperative Hypotension
Keywords: Intraoperative hypotension; Peripheral perfusion indexI; General anesthesia; Non-cardiac surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPI guided strategies (Experimental): The decision making for prevention and treatment of hypotension was PPI guided to maintain the PPI between 1 and 3.
  Interventions: Behavioral: PPI guided strategies
- conventional strategies (Other): The decision making for prevention and treatment of hypotension dependent on the experience of anesthesiologist.
  Interventions: Behavioral: Empirical strategies

INTERVENTIONS:
Behavioral: PPI guided strategies — For targeted MAP or lower, if PPI<1, more fluid therapy. if PPI>3, vasoconstriction therapy. For MAP<65mmHg and 1<=PPI<3, test bolus of 250 ml crystalloid fluid.
  Arms: PPI guided strategies
Behavioral: Empirical strategies — Fluid therapy or vasoconstriction depended on experiences of anesthetic staffs.
  Arms: conventional strategies

SUMMARY:
Intraoperative hypotension is closely related to the poor prognosis of surgery. The study is focused on the effectiveness of maintaining normal peripheral perfusion index (PPI) on time-weighted average of hypotension during anesthesia.

DETAILED DESCRIPTION:
Intraoperative hypotension is closely related to the poor prognosis of surgery. Hypotension decreased blood flow perfusion of organs, which lead to dysfunction of multiple organs, especially increasing serious complications such as cardio-cerebrovascular events and acute renal injury within 30 days after surgery. The aim of this study is to establish a set of strategies that can effectively prevent and treat intraoperative hypotension, so as to alleviate possible harm to patients from perioperative hypotension. The study is focused on the effectiveness of maintaining normal peripheral perfusion index (PPI) on time-weighted average of hypotension during anesthesia. The lower target mean arterial pressure (MAP) was higher than 65 mmHg. MAP less than 65 mmHg was defined as intraoperative hypotension between induction and tracheal extubation.

ELIGIBILITY:
Inclusion Criteria:

65 years and older ASA Physical Status 1-3 general anesthesia arterial catheterization procedures last more than 2 hours communicate normally in Mandarin

Exclusion Criteria:

abnormal Allen's test higher target than 65 mmHg history of diabetes vascular diseases arrhythmia cardiac function class II and above physical disability, unable to conduct PPI monitoring participated in other clinical studies in the past month

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
time-weighted average of hypotension (TWA)<65mmHg | Intraoperative (between anesthesia induction and tracheal extubation)
  total area under MAP<65 mmHg/surgery length

SECONDARY OUTCOMES:
Rate of hypotension after anesthesia induction | from anesthesia induction to 15 minutes after then
  the number of participants of hypotension/ the number of each group
Cumulative number of intraoperative hypotension episodes | Intraoperative (between anesthesia induction and tracheal extubation)
  Cumulative number of MAP<65mmHg and last at least for three minutes
Cumulative time of intraoperative hypotension period | Intraoperative (between anesthesia induction and tracheal extubation)
  Cumulative time of MAP<65mmHg
Proportion of time with hypotension | Intraoperative (between anesthesia induction and tracheal extubation)
  Proportion of cumulative time of intraoperative hypotension period and the anesthesia time
time-weighted average of hypertension (TWA)>100mmHg | Intraoperative (between anesthesia induction and tracheal extubation)
  total area under MAP>100 mmHg/surgery length
Cumulative number of intraoperative hypertension episodes | Intraoperative (between anesthesia induction and tracheal extubation)
  Cumulative number of MAP>100 mmHg and last at least for three minutes
postoperative plasma concentration of lactic acid | 5 minutes before and 5 minutes after the end of surgery
  Plasma concentration of lactic acid in the end of surgery
arterial partial pressure of oxygen (PaO2)/inspired fraction of oxygen (FiO2) | 5 minutes before and 5 minutes after the end of surgery
  PaO2/FiO2
intraoperative urine output | Intraoperative (between anesthesia induction and tracheal extubation)
  urine output during the surgery
the rate of acute kidney injury (AKI) | within 7 days after the end of surgery
  the number of participants with AKI/ the number of each group

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqiang Zhou, Principal Investigator — Tongji Hospital
Locations (1):
- Zhiqiang Zhou, Wuhan, China